CLINICAL TRIAL: NCT05687344
Title: Intensive Postpartum Antihypertensive Treatment to Improve Women's Cardiovascular Health (IPAT Study)
Brief Title: Intensive Postpartum Antihypertensive Treatment
Acronym: IPAT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Anna Palatnik, MD, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO00046214
Record Dates: First submitted 2023-01-01; First posted 2023-01-18 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Hypertensive Disorder of Pregnancy
MeSH Terms: conditions — Toxemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): Intervention group - intensive postpartum BP control with Nifedipine initiation at SBP≥140 mmHg or DBP≥90 mmHg and maintaining BP at <140/90 mmHg during the first 6 weeks postpartum. In addition, participants will receive education on healthy lifestyle following AHA LE8.
  Interventions: Drug: Nifedipine ER
- Active control arm (Active Comparator): Active control group - a group of usual care that follows ACOG recommendations with Nifedipine initiation at SBP≥150 mmHg or DBP≥100 mm Hg and maintaining BP at <150/100 mmHg during the first 6 weeks postpartum. In addition, participants will receive education on healthy lifestyle following AHA LE8.
  Interventions: Drug: Nifedipine ER

INTERVENTIONS:
Drug: Nifedipine ER — Postpartum BP treatment to <140/90 mmHg
  Other Names: Tight BP control group

SUMMARY:
The long-term goal of our work is to evaluate the effect of intensive postpartum blood pressure control on maternal cardiovascular health, risk of chronic hypertension, and reversal of vascular dysfunction generated by hypertensive disorders of pregnancy, thus attenuating the lifelong trajectory of cardiovascular disease risk.

DETAILED DESCRIPTION:
The IPAT will randomize 60 postpartum patients with HDP at the Medical College of Wisconsin (MCW) to intensive BP control with Nifedipine extended release (ER) (target BP <140/90 mmHg) versus usual care (target BP <150/100 mmHg). Oversampling of Black patients with HDP will be done to ensure they comprise 50% of study participants. Patients enrolled in both arms will undergo education on healthy lifestyle following AHA "Life's Essential 8" (LE8) of tobacco cessation, physical activity, healthy sleep, and healthy diet with detailed overview of DASH throughout the first year postpartum with monthly virtual educational session delivered by a registered dietician and a life coach. Assessment of LE8 CVH score will be done after delivery, 6 weeks postpartum, and 12 months postpartum. Participants will also undergo vascular function assessment: endothelial dysfunction with brachial artery flow mediated dilation (FMD), arterial stiffness with carotid-femoral pulse wave velocity (cfPWV) and anti-angiogenic and inflammatory CVD biomarker with soluble fms-like tyrosine kinase (sFlt-1), at baseline, 6 weeks, and 12 months postpartum. The primary outcome is feasibility of all study procedures, including recruitment, retention, and adherence. Secondary outcomes are change in BP, CVH score, FMD, PWV, and sFlt-1 from baseline to 12 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* HDP diagnosis (gestational hypertension or preeclampsia) according to ACOG guidelines
* Postpartum day 0-3 and prior to discharge
* Able to communicate in English or in Spanish
* Age 18 - 45

Exclusion Criteria:

* Pre-gestational hypertension
* Pre-gestational diabetes ( type 1 or type 2)
* Intent to transfer postpartum to an outside institution of the participating centers
* Known allergy to nifedipine or other significant contraindication to nifedipine
* Inability or unwillingness to provide informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility in randomization | 12 months postpartum
  Proportion of patients who enroll out of all approached, eligible patients.
Feasibility in recruitment | 12 months postpartum
  Number of patients successfully enrolled per month during the study.
Feasibility in retention | 12 months postpartum
  Proportion of enrolled patients who complete all study visits during the 12 months follow-up.
Contamination | 12 months postpartum
  Percent of patients following other antihypertensive treatment regimens.

SECONDARY OUTCOMES:
New stage I hypertension | 12 months postpartum
  BP of ≥130/80 mmHg
Life's Essential 8 cardiovascular health score (range 0-100) | 12 months postpartum
  The score will be calculated using American Heart Association application
Life's Simple 7 CVH (range 0-14) | 12 months postpartum
  Same metrics as LE8 excluding sleep
Flow-mediated dilation | 12 months postpartum
  Brachial artery flow-mediated dilation will assess endothelial dysfunction.
Serum biomarkers of CVD risk | 12 months postpartum
  Anti-angiogenic marker: Soluble fms-like tyrosine kinase (sFlt-1)
arterial stiffness | 12 months postpartum
  Carotid-femoral pulse wave velocity will assess arterial stiffness

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Palatnik A, Sunji N, Peterson Z, Ohlendorf J, Pan AY, Kulinski J. Intensive postpartum antihypertensive treatment (IPAT) and healthy lifestyle education: Study protocol for a pilot randomized controlled trial for patients with hypertensive disorders of pregnancy. Contemp Clin Trials. 2024 Dec;147:107710. doi: 10.1016/j.cct.2024.107710. Epub 2024 Oct 10. PMID 39395531